CLINICAL TRIAL: NCT02164461
Title: A Phase 1 Study Evaluating High Dose ADXS11-001 Treatment in Women With Carcinoma of the Cervix (ADXS001-07)
Brief Title: Axalimogene Filolisbac (ADXS11-001) High Dose in Women With Human Papillomavirus (HPV) + Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advaxis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Lm-LLO-E7-1401 (ADXS001-07)
Record Dates: First submitted 2014-06-13; First posted 2014-06-16 (Estimated); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2023-12

CONDITIONS: Effects of Immunotherapy; Metastatic/Recurrent Cervical Cancer; Cervical Adenocarcinoma; Cervical Adenosquamous Cell Carcinoma; Cervical Squamous Cell Carcinoma; Cervical Small Cell Carcinoma; Stage III Cervical Cancer; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
Keywords: Adenocarcinoma; Carcinoma; Carcinoma, Squamous Cell; Uterine Cervical Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Small Cell; Carcinoma, Adenosquamous; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Squamous Cell; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Uterine Cervical Diseases; Uterine Diseases; Genital Diseases, Female
MeSH Terms: conditions — Uterine Cervical Neoplasms; Adenocarcinoma; Carcinoma; Carcinoma, Squamous Cell; Small Cell Lung Carcinoma; Carcinoma, Small Cell; Carcinoma, Adenosquamous; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Neoplasms, Squamous Cell; Uterine Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms by Site; Uterine Cervical Diseases; Uterine Diseases; Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Axalimogene filolisbac 1x10^9 cfu (Experimental): Participants with persistent, metastatic, or recurrent carcinoma of the cervix who failed conventional therapy received axalimogene filolisbac at dose of 1x10^9 colony forming units (cfu) by intravenous infusion, over 60 minutes duration, every 3 weeks (Q3W) in repeating 12-week treatment cycles (Day 1 of Weeks 1, 4, 7, and 10 of each cycle) until a discontinuation criterion was met. Participants received a 7-day course of oral antibiotic therapy starting approximately 72 hours (Day 4) after each administration of axalimogene filolisbac. Antibiotic therapy consisted of trimethoprim (80 mg)/sulfamethoxazole (400 mg) tablets (Bactrim) or trimethoprim (160 mg)/ sulfamethoxazole (800 mg) tablets (Bactrim DS), administered 3 times during the 7 consecutive days or ampicillin 500 mg 4 times daily for 7 consecutive days for participants with sulfa allergy.
  Interventions: Biological: Axalimogene filolisbac
- Axalimogene filolisbac 5x10^9 cfu (Experimental): Participants with persistent, metastatic, or recurrent carcinoma of the cervix who failed conventional therapy received axalimogene filolisbac at dose of 5x10^9 cfu by intravenous infusion, over 60 minutes duration, Q3W in repeating 12-week treatment cycles (Day 1 of Weeks 1, 4, 7, and 10 of each cycle) until a discontinuation criterion was met. Participants received a 7-day course of oral antibiotic therapy starting approximately 72 hours (Day 4) after each administration of axalimogene filolisbac. Antibiotic therapy consisted of trimethoprim (80 mg)/sulfamethoxazole (400 mg) tablets (Bactrim) or trimethoprim (160 mg)/ sulfamethoxazole (800 mg) tablets (Bactrim DS), administered 3 times during the 7 consecutive days or ampicillin 500 mg 4 times daily for 7 consecutive days for participants with sulfa allergy.
  Interventions: Biological: Axalimogene filolisbac
- Axalimogene filolisbac 1x10^10 cfu (Experimental): Participants with persistent, metastatic, or recurrent carcinoma of the cervix who failed conventional therapy received axalimogene filolisbac at dose of 1x10^10 cfu by intravenous infusion, over 60 minutes duration, Q3W in repeating 12-week treatment cycles (Day 1 of Weeks 1, 4, 7, and 10 of each cycle) until a discontinuation criterion was met. Participants received a 7-day course of oral antibiotic therapy starting approximately 72 hours (Day 4) after each administration of axalimogene filolisbac. Antibiotic therapy consisted of trimethoprim (80 mg)/sulfamethoxazole (400 mg) tablets (Bactrim) or trimethoprim (160 mg)/ sulfamethoxazole (800 mg) tablets (Bactrim DS), administered 3 times during the 7 consecutive days or ampicillin 500 mg 4 times daily for 7 consecutive days for participants with sulfa allergy.
  Interventions: Biological: Axalimogene filolisbac

INTERVENTIONS:
Biological: Axalimogene filolisbac
  Other Names: ADXS11-001

SUMMARY:
To evaluate the tolerability and safety of axalimogene filolisbac 1 x 10^10 colony forming units (cfu) administered with prophylactic premedication in repeating 3-dose study cycles in women with persistent, metastatic, or recurrent squamous and non-squamous carcinoma, adenosquamous, or adenocarcinoma of the cervix. To evaluate tumor response and progression-free survival (PFS) by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).

DETAILED DESCRIPTION:
In this Phase 1, open-label, multicenter dose-escalation study, participants with persistent, metastatic, or recurrent carcinoma of the cervix who failed conventional therapy received axalimogene filolisbac every 3 weeks in repeating 12-week treatment cycles. Axalimogene filolisbac was administered intravenously (IV) on Day 1 of Weeks 1, 4, 7, and 10 of each cycle. Participants received a prophylactic regimen that was completed prior to each axalimogene filolisbac infusion to mitigate and manage potential immune responses seen with immunotherapy administration. The pretreatment prophylaxis regimen included commercially available antihistamines, nonsteroidal anti-inflammatory drugs (NSAIDs), antiemetics, histamine H2-receptor antagonists, and IV hydration. Additional NSAID doses and antiemetic administration were given post initial administration on Day 1 and Day 2, at the discretion of the investigator.

Participants received a 7-day course of oral antibiotic therapy starting approximately 72 hours (Day 4) after each administration of axalimogene filolisbac. Antibiotic therapy consisted of trimethoprim (80 mg)/sulfamethoxazole (400 mg) tablets (Bactrim) or trimethoprim (160 mg)/ sulfamethoxazole (800 mg) tablets (Bactrim DS), administered 3 times during the 7 consecutive days or ampicillin 500 mg 4 times daily for 7 consecutive days for participants with sulfa allergy.

Axalimogene filolisbac doses were to be escalated/de-escalated in the standard 3 + 3 fashion, starting with 5x10^9 cfu to a maximum dose level of 1x10^10 cfu. Dose cohorts of 3 participants each were to be treated. All decisions regarding dose escalation/de-escalation were made by the sponsor in consultation with investigators. In the absence of dose-limiting toxicity (DLT) assessed during the first 28 days in Cycle 1, the dose was to be escalated to the next dose level for the next 3 participants. If DLT was seen in 1 of 3 participants, another 3 participants were to be treated at that same dose. If DLT was seen in 2 of 6 participants, then that dose level was considered the Maximum Tolerated Dose (MTD) and the previous dose level was selected as the Recommended Phase 2 dose (RP2D). Specific hematologic and non-hematologic DLT criteria were prospectively defined in protocol. The RP2D was to be selected based on an observed DLT rate of <33%.

Additional participants were to be enrolled into an expansion cohort to allow approximately 15 participants to be treated at that dose level.

Treatment cycles were repeated at the RP2D (or less) for an individual participant until a discontinuation criterion was met. Discontinuation criteria included documented disease progression, intolerable side effects not resolved with dose reduction or change in premedication or the participant completed 1 cycle of treatment post observation of complete response (CR per RECIST 1.1 and immune-realted complete response [irCR] per irRECIST). Participants who experienced a DLT during the dose-escalation portion of the study or experienced events meeting the definition of a DLT as described in the protocol in any subsequent treatment cycle were to be discontinued from study treatment. However, if a participant who experienced a DLT showed significant response to axalimogene filolisbac, the participant could receive subsequent axalimogene filolisbac treatment at a lower dose level following discussion and agreement between the investigator and sponsor.

Efficacy was assessed by tumor imaging at the end of every cycle. Safety was assessed by analyzing treatment-related adverse events (AEs), changes in physical examinations, vital sign measurements, and clinical laboratory abnormalities. All toxicities were graded using Common Terminology Criteria for Adverse Events (CTCAE) 4.03.

After the study treatment period, all participants were to participate in a 3-year Lm surveillance monitoring period that included a 6-month course of antibiotics to be initiated 72 hours after completion of treatment or immediately following study discontinuation and monitoring (Complete blood count [CBC], comprehensive metabolic panel, and blood cultures for the detection of Lm) every 3 months (±2 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically-confirmed, persistent, metastatic or recurrent squamous or non-squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix with documented disease progression (disease not amenable to surgery or standard radiotherapy).
* Participants who have received no more than 1 prior cytotoxic treatment regimen.
* Participant may have received ≤2 prior regimens for the treatment of their metastatic disease.
* Participant is able to provide written informed consent.
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* In the opinion of the investigator, participant has rapidly progressing disease, OR has life expectancy of less than 6 months, OR would be unable to receive at least one cycle of therapy.
* Participant has received chemotherapy and/or radiation therapy (except palliative radiation therapy for disease-related pain) within ≤2 weeks of first axalimogene filolisbac infusion.
* Participant has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has a contraindication to administration of trimethoprim/sulfamethoxazole or ampicillin.
* Has implanted medical device(s) that pose a high risk for colonization and/or cannot be easily removed (e.g., prosthetic joints, artificial heart valves, pacemakers, orthopedic screw(s), metal plate(s), bone graft(s), or other exogenous implant(s). NOTE: More common devices and prosthetics which include arterial and venous stents, dental and breast implants, and venous access devices (e.g., Port-a-Cath or Mediport) are permitted. Sponsor must be contacted prior to consenting any participant who has any other device and/or implant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Augusta, Georgia
  - Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with persistent, metastatic, or recurrent carcinoma of the cervix who failed conventional therapy were enrolled in this study.
Pre-assignment Details: Participants received a prophylactic regimen that was completed prior to each axalimogene filolisbac infusion to mitigate and manage potential immune responses seen with immunotherapy administration.
Period: Overall Study
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Started | 1 | 6 | 5
Enrolled Participants | 0 | 6 | 6
Treated Participants | 1 (one participant who was enrolled in the high-dose group received 1x10^9 cfu.) | 6 | 5
Completed | 0 | 0 | 0
Not Completed | 1 | 6 | 5
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Disease Progression | 1 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The All Treated population included participants who received at least 1 dose of study drug.
Groups:
- Axalimogene Filolisbac 1x10^9 Cfu: Participants with persistent, metastatic, or recurrent carcinoma of the cervix who failed conventional therapy received axalimogene filolisbac at dose of 1x10^9 cfu by intravenous infusion, over 60 minutes duration, Q3W in repeating 12-week treatment cycles (Day 1 of Weeks 1, 4, 7, and 10 of each cycle) until a discontinuation criterion was met. Participants received a 7-day course of oral antibiotic therapy starting approximately 72 hours (Day 4) after each administration of axalimogene filolisbac. Antibiotic therapy consisted of trimethoprim (80 mg)/sulfamethoxazole (400 mg) tablets (Bactrim) or trimethoprim (160 mg)/ sulfamethoxazole (800 mg) tablets (Bactrim DS), administered 3 times during the 7 consecutive days or ampicillin 500 mg 4 times daily for 7 consecutive days for participants with sulfa allergy.
- Total: Total of all reporting groups
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu | Total
Number analyzed (Participants) | 1 | 6 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 | 51.3 (11.22) | 59.2 (19.10) | 53.6 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 5 | 12
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 6 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 3 | 5
  White | 1 | 4 | 2 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as occurrence of any of the following toxicities that are possibly, probably or definitely related to therapy.
  Hematologic:
  1. Grade 4 hematologic toxicity.
  2. Febrile neutropenia, defined as absolute neutrophil count (ANC) < 1000/mm^3 with a single temperature of >38.3° C (101° F) or a sustained temperature of >38° C (100.4° F) for more than 1 hour.
  3. Grade 3 thrombocytopenia lasting >72 hours.
  4. Grade 4 thrombocytopenia.
  Non-Hematologic:
  1. ≥Grade 3 non-hematologic toxicity
  2. Grade 3 non hematologic laboratory values.
  3. Listeremia: positive blood cultures along with persistent (for 72 hours post dose) symptoms consistent with listeremia (e.g., fever and muscle aches, often preceded by diarrhea or other gastrointestinal symptoms).
  4. ≥Grade 3 flu-like symptoms or cytokine release symptoms that persist for >24 hours after study treatment administration despite symptomatic treatment.
Time Frame: Up to 28 days in Cycle 1 (12 weeks cycle)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
Participants | 0 | 1 | 0

2. Primary Outcome: Listeria Monocytogenes Surveillance
Description: Number of participants with delayed listeria infection was reported.
Time Frame: Up to 120 days post dose
Population: All Treated Participants
Measure: Number; unit: participants
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse event (AE): any untoward medical occurrence in a participant administered a study treatment & which did not necessarily have to have a causal relationship with the study treatment. An AE is, any unfavorable & unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of study treatment. AE with onset on or after the date of first administration of the study treatment until the end of the Listeria Monocytogenes (Lm) surveillance period.
Time Frame: From first dose up to 2.3 years
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
Participants | 1 | 6 | 5

4. Secondary Outcome: Objective Response Rate (ORR) as Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: ORR as per RECIST 1.1 was defined as the percentage of participants who achieved complete response (CR) or partial response (PR). CR was defined as disappearance of all lesions. PR was defined as ≥30% decrease in the sum of the longest diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: From first dose until end of treatment (Maximum duration: 1.5 years)
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
percentage of participants | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93] | 20.00 [0.51 to 71.64]

5. Secondary Outcome: Duration of Tumor Response as Per RECIST 1.1
Description: Duration of response as per RECIST 1.1 was defined as the time interval from CR or PR to disease progression or death. CR was defined as disappearance of all lesions. PR was defined as ≥30% decrease in the sum of the longest diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Progressive disease (PD) was defined as at least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of one or more new lesions is also considered progression .Kaplan-Meier method was used to estimate median and 95% confidence interval (CI).
Time Frame: From first objective response to disease progression or death (Maximum duration: 1.5 years)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
days | NA [NA to NA] — Median and 95% CI was not estimable as there were no events | NA [NA to NA] — Median and 95% CI was not estimable as there were no events | 269.0 [NA to NA] — 95% CI was not estimable due to low number of events

6. Secondary Outcome: Progression Free Survival (PFS) as Per RECIST 1.1
Description: PFS as per RECIST 1.1 was defined as the time interval from study enrollment to disease progression or death. Participants who were alive with no disease progression were censored at the date of the last tumor assessment. PD was defined as at least 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. The appearance of one or more new lesions is also considered progression.The Kaplan-Meier method was used to estimate median and 95% CI.
Time Frame: From study enrollment to disease progression or death (Maximum duration: 1.5 years)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
days | 124.0 [NA to NA] — 95% CI was not estimable due to low number of events | 85.0 [80.0 to 99.0] | 176.5 [78.0 to 528.0]

7. Secondary Outcome: ORR as Per Immune-related Response Evaluation Criteria in Solid Tumors (irRECIST)
Description: ORR as per irRECIST was defined as the percent of participants who achieved immune response complete response (irCR) or immune response partial response (irPR). irCR was defined as disappearance of all lesions. irPR was defined as ≥30% decrease in tumor burden compared with baseline.
Time Frame: From first dose until end of treatment (Maximum duration was 1.5 years)
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
percentage of participants | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 45.93] | 20.00 [0.51 to 71.64]

8. Secondary Outcome: Duration of Tumor Response as Per irRECIST
Description: Duration of response as per irRECIST 1.1 was defined as the time interval from irCR or irPR to disease progression or death. irCR was defined as disappearance of all lesions. irPR was defined as ≥30% decrease in tumor burden compared with baseline. Immune response progressive disease (irPD) was defined as at least 20% increase in tumor burden compared with nadir (at any single time point). The Kaplan-Meier method was used to estimate median and 95% CI.
Time Frame: From first objective response to disease progression or death (Maximum duration: 1.5 years)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
days | NA [NA to NA] — Median and 95% CI was not estimable as there were no events | NA [NA to NA] — Median and 95% CI was not estimable as there were no events | 269.0 [NA to NA] — 95% CI was not estimable due to low number of events

9. Secondary Outcome: PFS as Per irRECIST
Description: PFS as per irRECIST 1.1 was defined as the time interval from study enrollment to disease progression or death. Participants who were alive with no disease progression were censored at the date of the last tumor assessment. irPD was defined as at least 20% increase in tumor burden compared with nadir (at any single time point). The Kaplan-Meier method was used to estimate median and 95% CI.
Time Frame: From study enrollment to disease progression or death (Maximum duration: 1.5 years)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
Number analyzed (Participants) | 1 | 6 | 5
days | 124.0 [NA to NA] — 95% CI was not estimable due to low number of events | 85.0 [80.0 to 99.0] | 176.5 [78.0 to 528.0]

ADVERSE EVENTS:
Time Frame: 2 years and 3 days.
Description: All Treated Participants
Arm/Group | Axalimogene Filolisbac 1x10^9 Cfu | Axalimogene Filolisbac 5x10^9 Cfu | Axalimogene Filolisbac 1x10^10 Cfu
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/6 | 2/5
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/6 | 1/5
Other Adverse Events (participants affected / at risk) | 1/1 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axalimogene Filolisbac 1x10^9 Cfu (N=1) | Axalimogene Filolisbac 5x10^9 Cfu (N=6) | Axalimogene Filolisbac 1x10^10 Cfu (N=5)
Hypotension (Vascular disorders) | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axalimogene Filolisbac 1x10^9 Cfu (N=1) | Axalimogene Filolisbac 5x10^9 Cfu (N=6) | Axalimogene Filolisbac 1x10^10 Cfu (N=5)
Tachycardia (Cardiac disorders) | 1 | 2 | 2
Pyrexia (General disorders) | 1 | 2 | 4
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 4 | 3
Malaise (General disorders) | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 1
Capillary nail refill test abnormal (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Skin turgor decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2
Aura (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 2
Catheter site pain (General disorders) | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1
Listeria test positive (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall seek the Sponsor's written approval for study results publication which shall not be unreasonably withheld. Such publication by Institution and/or Investigator may be no earlier than after a cooperative publication has been published with Sponsor or 1 year from date of completion or termination of the Study & only after review and comment by Sponsor. Institution agrees to provide Sponsor a copy of proposed publication at least 60 days prior to submission to a publisher.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT02164461/Prot_SAP_000.pdf